CLINICAL TRIAL: NCT04288349
Title: Intraoperative Use of Perineal Block for Hemorrhoidectomy
Acronym: IREN
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Russian Society of Colorectal Surgeons (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1
Record Dates: First submitted 2020-02-26; First posted 2020-02-28 (Actual); Last update posted 2020-05-29 (Actual); Status verified 2020-05

CONDITIONS: Hemorrhoidectomy; Pudendal Nerve
Keywords: perineal block; hemorrhoidectomy; hemorrhoids; hemorrhoids treatment; pudendal nerve
MeSH Terms: conditions — Hemorrhoids | interventions — Epinephrine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Randomization of the patients included in the study was performed before surgery. Patients were being randomly divided into two groups. All patients getting subarachnoid anesthesia. Perineal block using solution of ropivocaine and epinephrine for the first group was performed and placebo with epinephrine - for the second group. A researcher who does not participate in the surgery and does not contact with patients at all perioperative stages performs randomization and prepares a solution block. Neither the patient nor the operating surgeon and the doctors who register the results of the treatment are not informed about the anesthesia used in each case.
  The probability of introduction to each group is 50%. The number of patients in both groups equally and is 50 people.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- epinephrine + ropivacaine +saline (Active Comparator): 1% epinephrine solution + 30 ml of 1% ropivacaine solution diluted with 20 ml of 0.9% saline for achievement a 0.75% anesthetic solution in a ratio of 1: 200 000
  Interventions: Procedure: perineal block with usage of one of solutions; Drug: epinephrine + ropivacaine +saline
- epinephrine + saline (Placebo Comparator): 1% epinephrine solution + 50 ml of 0.9% saline in a ratio of 1: 200 000.
  Interventions: Procedure: perineal block with usage of one of solutions; Drug: epinephrine + saline

INTERVENTIONS:
Procedure: perineal block with usage of one of solutions — Perineal block using solution of ropivocaine and epinephrine for the first group was performed. Anococcygeal ligament is infiltrated with 10 ml of the solution after the intracutaneous infiltration in 2 cm from the anus. Ten ml of the solution is injected in ischiorectal fat on each side. The needle is orienteered at the angle of 45 degrees cranially and laterally, and to the surface what allows the surgeon to anesthetize the deep branches of the pudendal nerve. In addition, 10 ml of solution is injected transdermal on the front edge of the anus with further subcutaneous infiltration on each side of the anus to provide anesthesia to the nerve branches laying more superficial. The total amount of the injected solution is 50 ml.
Drug: epinephrine + ropivacaine +saline — epinephrine + ropivacaine +saline
  Arms: epinephrine + ropivacaine +saline
Drug: epinephrine + saline — epinephrine + saline
  Arms: epinephrine + saline

SUMMARY:
Perineal block with the anesthesia of the pudendal nerve's terminal branches allows to perform a hemorrhoidectomy with the optimal intraoperative and postoperative analgesia The purpose of this study is to assess the effectiveness of the intraoperative use of perineal block with spinal anesthesia to reduce postoperative pain and the amount of used analgesics.

DETAILED DESCRIPTION:
Hemorrhoidectomy, as has being demonstrated to be an effective method of treatment for stage III-IV hemorrhoidal disease. However it is associated with intense postoperative pain that requires the use of multimodal analgesia. Inadequate pain control leads to the prolongation of admission, increasing the consumption of opioid analgesics.

Traditionally spinal or general anesthesia is used in proctological practice. However, the number of studies about using of perianal local anesthesia, both in combination with general anesthesia and as a separate practice has been increasing recently.

Perineal block with the anesthesia of the pudendal nerve's terminal branches allows to perform a hemorrhoidectomy with the optimal intraoperative and postoperative analgesia. The drugs used for this have some pharmacological differences in the duration of the drug and the form of administration.

The aim of this prospective, randomized, double-blind study is to assess the effectiveness of the intraoperative use of perineal block with spinal anesthesia to reduce postoperative pain and the amount of used analgesics.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent.
2. Patients over 18 years.
3. Symptomatic grade III-IV hemorrhoids.
4. Planned surgery: Milligan-Morgan hemorrhoidectomy.

Exclusion Criteria:

1. Patient's refuse to participate in the study.
2. Pregnancy.
3. Сontraindications or technical inability to perform subarachnoid anesthesia.
4. Decompensated somatic diseases.
5. Inflammation of the perianal region.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-02-20 (Actual); Primary Completion 2020-05-29 (Estimated); Study Completion 2020-05-30 (Estimated)

PRIMARY OUTCOMES:
The rate of opioid analgesics usage | 1 day - 2 weeks
  The need to use opioid analgesics.

SECONDARY OUTCOMES:
systemic analgesics usage | 1 day - 2 weeks
  The duration and frequency of systemic analgesics usage, including opioid and topical local anesthetics in early postoperative period. The assessment of the required amount and frequency of NSAIDs (nonsteroidal anti-inflammatory drugs) usage in the first 24 hours, then - daily up to 7 days
The duration of painless period after surgery | 1 day - 1 week
  the time from the moment of the blockade to the need of intake the first dose of analgesics.
re-admission | 1 day - 1 month
  The need for re-admission after operation
quality of life with SF-36 questionnaire | 1 day - 1 month
  The assessment of quality of life after surgery using the SF-36 questionnaire (The Short Form-36). Scale evaluates physical and mental status after operation.
The timing of returning to work. | 1 day - 1 month
  The period between surgery and returning to normal work
early postoperative complications | 1 day - 1 month
  Assessment of early postoperative complications (bleeding, retention of urine, infectious complications).

CONTACTS AND LOCATIONS:
Overall Officials: Petr Tsarkov, Prof, Principal Investigator — Russian Society of Colorectal Surgeons
Locations (1):
- Clinic of Colorectal and Minimally Invasive Surgery, Moscow, Russia